CLINICAL TRIAL: NCT04595422
Title: Educating Smokers About Lung Cancer Screening Using Tobacco Quitlines
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2020-0013; NCI-2020-03812 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2020-0013 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2020-07-15; First posted 2020-10-20 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-10

CONDITIONS: Lung Carcinoma
MeSH Terms: conditions — Lung Neoplasms | interventions — Early Intervention, Educational; Educational Status; Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Call center staff (educational intervention) (Experimental): Participants undergo training consisting of a 60-minute educational session.
  Interventions: Other: Educational Intervention; Other: Survey Administration
- Callers substudy (LCS educational materials, questionnaire) (Experimental): Participants are referred to lung cancer screening educational materials. Participants also complete questionnaires at 1 week and 6 months after referral to educational materials.
  Interventions: Other: Educational Intervention; Other: Questionnaire Administration

INTERVENTIONS:
Other: Educational Intervention — Undergo training consisting of a 60-minute educational session
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Call center staff (educational intervention)
Other: Educational Intervention — Receive lung cancer screening educational materials
  Other Names: Education for Intervention; Intervention by Education; Intervention through Education; Intervention, Educational
  Arms: Callers substudy (LCS educational materials, questionnaire)
Other: Questionnaire Administration — Complete questionnaire
  Arms: Callers substudy (LCS educational materials, questionnaire)
Other: Survey Administration — Ancillary studies
  Arms: Call center staff (educational intervention)

SUMMARY:
This implementation study will examine the best ways to refer heavy smokers to information about lung cancer screening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To increase the number of smokers eligible for lung cancer screening (LCS) who receive high-quality educational materials about LCS through tobacco quitlines.

OUTLINE:

CALL CENTER STAFF: Participants undergo training consisting of a 60-minute educational session.

CALLERS SUBSTUDY: Participants are referred to lung cancer screening educational materials. Participants also complete questionnaires at 1 week and 6 months after referral to educational materials.

ELIGIBILITY:
Inclusion Criteria:

* QUITLINE CALL CENTER STAFF
* Staff member of a quitline
* Aged 18 years and above
* CALLERS (SMOKERS WHO CONTACT THE QUITLINE ABOUT SMOKING CESSATION SERVICES) INCLUSION CRITERIA
* Callers 55-80 years of age
* Current smoker, or former smoker with a cessation history of < 15 years
* >= 30 pack-year smoking history
* English-speaking

Exclusion Criteria:

* CALLERS (SMOKERS WHO CONTACT THE QUITLINE ABOUT SMOKING CESSATION SERVICES) EXCLUSION CRITERIA
* History of lung cancer by self-report

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2020-07-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Content from communications (email, phone, monthly calls) | Up to 4 years
  Will be content analyzed using Atlas.ti qualitative software according to the adaptation framework from Stirman and colleagues. Will identify 1) who made the modification; 2) what was modified (i.e., content, context, training and evaluation); 3) for whom the modification was made (e.g., individual counselor); 4) context of the modification (e.g., format, setting, personnel, population); and 5) what was the nature of the modification (e.g., adding elements). Will also code for facilitators and barriers that are consistent with the constructs from CFIR. All textual data will be double coded and discussed by the researchers.
Healthcare sector perspective | Up to 4 years
  As needed, will use a process-flow analysis to identify all resources utilized at each of the step of the program.
Reach | During 6 month implementation period
  The analysis of the data from the logs and surveys will include examining the means, medians, standard deviations, and ranges overall and by state quitline for Reach
Overall lung cancer screening rate | Up to 6 months
Effectiveness (Caller Substudy) | Up to 6 months
  Will be successful if callers who participate in the evaluation answer at least 58 percent (7/12) of the Adapted lung cancer screening (LCS)-12 Knowledge Measure questions correctly and have a PrepDM score of at least 80 (standard deviation [SD] = 17.7), which were observed in the original project.

CONTACTS AND LOCATIONS:
Overall Officials: Robert J Volk, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M D Anderson Cancer Center — http://www.mdanderson.org